CLINICAL TRIAL: NCT01452893
Title: Counterregulatory Hormone Production and Cognitive Function in Patients With Adrenal Insufficiency and Diabetes Mellitus Type I
Brief Title: Counterregulatory Hormone Production in Adrenal Insufficiency and Diabetes Type I
Acronym: CANDI
Status: Completed | Type: Observational
Sponsor: University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Bruno Allolio, professor of medicine, head of the department of endocrinology and diabetology, University of Wuerzburg
Other Study IDs: CANDI-1
Record Dates: First submitted 2011-09-29; First posted 2011-10-17 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Addison's Disease; Adrenal Insufficiency; Diabetes Mellitus Type I
MeSH Terms: conditions — Addison Disease; Adrenal Insufficiency; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for hormonal analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Type I diabetes: Adult patients with diabetes mellitus type I but normal adrenal function
  Interventions: Procedure: Spiroergometry
- Addison's disease: Adult patients with Addison's disease
  Interventions: Procedure: Spiroergometry
- Type I diabetes and Addison's disease: Patients suffering from both, diabetes mellitus type I and Addison's disease
  Interventions: Procedure: Spiroergometry
- healthy controls: healthy controls with normal adrenal function and normal glucose regulation
  Interventions: Procedure: Spiroergometry

INTERVENTIONS:
Procedure: Spiroergometry — At visit 1 determination of the individual VO2max (maximal oxygen uptake) by spiroergometry after first testing of cognitive function.
  At visit 2: Spiroergometry with 3 min warm up followed by 5 min 50% VO2max and 15 min at the individual respiratory compensation point (RCP).

SUMMARY:
Patients with adrenal insufficiency also exhibit an adrenomedullary dysfunction. Furthermore, patients who suffer from both, adrenal insufficiency and type I diabetes more frequently report hypoglycemia, particularly after strenuous activities. The study investigates the counter regulatory hormonal response to physical stress and the impact on cognitive function in subjects with and without Addison's disease, type I diabetes and healthy subjects.

DETAILED DESCRIPTION:
As patients with adrenal insufficiency also exhibit an adrenomedullary dysfunction and patients who suffer from both, adrenal insufficiency and type I diabetes more frequently report hypoglycemia, particularly after strenuous activities this study investigates the counter-regulatory hormonal response to physical stress and the impact on cognitive function in subjects with and without Addison's disease, type I diabetes and healthy subjects. Patients will perform ergometer training with an individualized intensity and fulfill cognitive function testing (stroop test and fatigue inventories) before and after strenuous activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Addison's disease and/or diabetes mellitus type I or healthy control with normal adrenal function and normal glucose regulation
* Age ≥ 18 years
* Ability to comply with the study protocol
* Capability to perform spiroergometry

Exclusion Criteria:

* Any contraindication for performing spiroergometry according to the guidelines of the German Cardiac Society:

  * acute myocardial infarction
  * instable angina pectoris
  * symptomatic arrhythmia
  * severe and symptomatic stenosis of the aortic valve
  * decompensated heart failure
  * acute pulmonary embolism
  * Acute myocarditis
  * Acute pericarditis
  * Acute aortic dissection
  * main coronary artery disease
  * valvulopathies
  * electrolyte disturbance
  * arterial hypertension (systolic blood pressure > 200 mm Hg, diastolic BP > 110 mm Hg)
  * Tachyarrhythmia or Bradyarrhythmia
  * Hypertrophic cardiomyopathy and other forms of obstructive heart disease
  * second or third degree atrioventricular block
* Fever
* Diabetes mellitus Type 2
* Diseases or medication influencing the endogenous levels of plasma catecholamines(e. g. pheochromocytoma, paraganglioma, antidepressants, levodopa)
* Glucocorticoid-pharmacotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Four groups:
  Patients with Addison's disease alone patients with diabetes mellitus type I alone patients with both, Addison's disease and Diabetes mellitus type I healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
difference in cognitive function before and after physical stress | testing is performed at first visit (baseline, duration 5 min) and second visit (at least 48 hours after visit1). The second test is performed 5 min after strenous activity of 23 min duration, test duration again 5 min)
  study participants are tested with three standardized tests: stroop-task, symptom rating scale and a short term memory test. First testing is performed at visit 1 at rest, the second test at visit 2 after strenuous activity at a bicycle ergometer.

SECONDARY OUTCOMES:
differences in counterregulatory hormonal response to physical stress | at visit 2, blood sampling over 180 min starting 10 min before spiroergometry
  blood samples for determination of blood glucose, catecholamines and other counterregulatory hormones (cortisol, growth hormone) are collected before, during and after physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Allolio, MD, Study Chair — University of Wuerzburg; Stefanie Hahner, MD, Principal Investigator — University of Wuerzburg
Locations (1):
- Dept. of Endocrinology and Diabetology, Dept. of Medicine I, University Hospital Wuerzburg, Würzburg, Germany